CLINICAL TRIAL: NCT05157802
Title: Promoting Physical Activity Engagement for People With Early-stage Cerebellar Ataxia (EngageAtaxia)
Brief Title: Promoting Physical Activity Engagement for People With Early-stage Cerebellar Ataxia
Acronym: EngageAtaxia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-042
Record Dates: First submitted 2021-11-24; First posted 2021-12-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cerebellar Ataxia
Keywords: physical activity; physical therapy; balance training; physical activity coaching; neurodegenerative disease; rehabilitation
MeSH Terms: conditions — Cerebellar Ataxia; Motor Activity; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Coaching (Experimental): Participants will receive up to 5 individualized coaching sessions delivered via telehealth to facilitate and optimize exercise uptake. The therapist will facilitate discussion on specific and measurable goals, and will provide options for tracking their progress, such as written or web-based exercise logs or an activity monitor. The recommended exercises will be individualized to each participant but will primarily focus on increasing general physical activity (e.g. steps per day) as well as engagement in moderate intensity aerobic exercise a minimum of three times per week. Balance and strengthening exercises will also be recommended as appropriate.
  Interventions: Behavioral: Physical activity coaching

INTERVENTIONS:
Behavioral: Physical activity coaching — Physical activity coaching over 5 sessions

SUMMARY:
Engage-Ataxia will implement a physical activity coaching program for people with cerebellar ataxia at Teachers College, Columbia University. This program expands upon the current Engage program for people with Parkinson's disease (Engage-PD), an exercise coaching program for people with early stage Parkinson's disease to target individuals with early stage cerebellar ataxia. Engage-Ataxia will utilize a physical or occupational therapist to provide up to five one-on-one coaching sessions for individuals newly diagnosed with cerebellar ataxia. Therapists will work with participants to provide individualized structured support to facilitate and optimize exercise uptake as one part of comprehensive disease management. Participants will undertake two assessments three months apart, and will receive coaching interventions via Zoom healthcare platform. The primary objective of this program is to increase physical activity and exercise engagement in individuals with early stage cerebellar ataxia. This feasibility study will provide preliminary data and insight into the benefits of a remote coaching intervention for people with cerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist confirmed diagnosis of cerebellar ataxia
* Scale for Ataxia Rating and Assessment (SARA) score between 8-25 (total score of 40), which will capture mild to moderate stage of the disease
* Ambulatory for indoor and outdoor mobility without assistance or assistive device
* Successful completion of Physical Activity Readiness Questionnaire (PAR-Q) or medical clearance from primary doctor
* Medical clearance to exercise

Exclusion Criteria:

* Musculoskeletal injury that would prevent participation in an exercise program
* Other neurological disease or disorder such as stroke
* Cardiac/pulmonary conditions that would affect participants ability to participate exercise program
* Metabolic conditions that would affect participants during an exercise program
* Currently do moderate-vigorous exercise 5 days a week or more

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Scale for Assessment and Rating for Ataxia | Baseline, Post-Intervention (3 months)
  Clinical rating scale for severity of ataxia symptoms. This is an 8-item clinical performance based scale, which individuals are graded according to total ataxia severity. Total scores can range from 0 (no ataxia) to 40 (most severe ataxia). Scores are based on performance of the following tasks: 1) Gait, 2) Stance, 3), Sitting, 4) Speech Disturbance, 5) Finger Chase, 6) Nose-Finger Test, 7) Fast alternating hand movements, 8) Heel-shin slide. For the purpose of this study, we will be performing a modified version of the SARA, and be using the first four items of the SARA Scale (Gait, Stance, Walking, Speech) to be administered via telehealth.
Change in Cerebellar Cognitive Affective Syndrome Scale | Baseline, Post-Intervention (3 months)
  The Cerebellar Cognitive Affective Syndrome Scale (CCAS) was developed as a bedside quick screen for Cerebellar Cognitive Affective Symptom (also referred to as Schmalmann's Syndrome). The CCAS is a 10-item scale of cognitive and neuropsychiatric tests detailing executive function, working and verbal memory, language, visuospatial function, abstract reasoning, behavior and affect. Two scores are reported; a raw score ranging from 0 (severe cognitive impairment) to 120 points (no cognitive impairment), as well as a Pass/Fail marker for each of the 10 items on the scale. 1 fail is considered as possible cerebellar cognitive affective symptom, 2 fails are considered probable, and 3 fails are considered clinically definite.
Change in Brunel Lifestyle Physical Activity Questionnaire | Baseline, Post-Intervention (3 months)
  Evaluates both pre-planned and unplanned physical activity. Both pre-planned and unplanned physical activity subsections are separately scored through summation and average. Higher averages (closer to 5) indicate greater physical activity, whereas lower averages (closer to 0) indicate little to no physical activity in either category.

SECONDARY OUTCOMES:
Exercise Identity Scale Exercise Identity Scale | Baseline, Post-Intervention (3 months)
  Questions pertaining to salience of exercise identity. Scores range from 0 (no exercise identity) to 45 (high degree of exercise identity).
The Self- Efficacy for Exercise Scale | Baseline, Post-Intervention (3 months)
  Assesses an individual's beliefs in their ability to engage with exercise. Scores range from 0 (no exercise self-efficacy) to 90 (high exercise self efficacy).
Activities Specific Balance Scale (ABC) | Baseline, Post-Intervention (3 months)
  This assessment is a patient reported outcome evaluating the balance confidence of a participant in performing a variety of activities without losing balance or experiencing a state of unsteadiness. Participants are asked to rank their perceived balance confidence on a scale of 0% (no balance confidence) to 100% (high balance confidence). All scores are summed, and averaged for a total overall estimate of balance confidence.
Digital Biomarker of Static Posturography | Baseline, Post-Intervention (3 months)
  Participant will perform static standing with feet together and postural sway will be recorded with a smart phone app.
Digital Biomarker of Dynamic Posturography | Baseline, Post-Intervention (3 months)
  Participant will perform the Timed Up and Go Test (TUG) which consists of standing from a seated position, walking forward 10 feet, turning around, walking back 10 feet, and then returning to a seated position. The TUG test will be recorded with a smart phone app.
Acceptability Questionnaire | Post-intervention (3 months)
  A short open-ended questionnaire to assess the acceptability of the intervention. These open-ended questions will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No